CLINICAL TRIAL: NCT01561170
Title: The Effect of Electromagnetic Field Therapy to Improve Healing of Chronically Venous Ulcer in Lower Extremities
Brief Title: Electromagnetic Field Therapy to Improve Healing of Chronically Venous Ulcer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: N-20110052
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Venous Hypertension With Ulcer and Inflammation; Venous Ulcer Pain
Keywords: Electromagnetic; Field therapy; Chronically venous ulcer; Venous insufficiens
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronically venous ulcer: A group of 36 patients
  Interventions: Device: Active Pulsed Electro-Magnetic Field (PEMF); Device: Placebo Pulsed Electro-Magnetic Field (PEMF)

INTERVENTIONS:
Device: Active Pulsed Electro-Magnetic Field (PEMF) — One group of patients receive active devices. Both patients and investigator are blinded.
  Other Names: No other names.
Device: Placebo Pulsed Electro-Magnetic Field (PEMF) — One group of patients receive placebo devices. Both patients and investigator are blinded.
  Other Names: No other names.

SUMMARY:
Chronically venous ulcer in lower extremities is a permanent and disabling disease. Venous insufficience is the main cause of chronic ulcer. There is a high prevalence and frequency of the disease, primarily among elderly people. Recently, electromagnetic field therapy has been tested on various diseases in musculoskeletal system with a beneficial effect. In recent years, there has been an increasing interest in using electromagnetic field therapy to treat chronically venous ulcer.

The hypothesis of the investigators is that the electronic magnetic field therapy improves the healing process and reduces pain for patients suffering from chronically venous ulcer. The investigators assume that the bioactivity is affected by a cellular response which affects the DNA synthesis, transcription og protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from ulcer in lower extremities
* Patients who suffer from venous insufficience detected by duplex scanning or by a pressure on digits > 40 mmHg
* Patients with a regular need of compression stockings
* Age > 18 years

Exclusion Criteria:

* Age < 18 years
* Unability to read or understand Danish
* Patients who suffer from manifest neoplastic disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of ulcerous area. | 3 months
  Measurement of ulcerous area in order to assessing the effect of the healing process.

SECONDARY OUTCOMES:
Pain reduction in proportion to Visual Analogue Scale (VAS). | 3 months
  The pain reduction will be measured by VAS and an analysis of the medication between the two group of patients will be carried out in order to measure quality of life, adverse effects, ulceration, granulation tissue etc.

CONTACTS AND LOCATIONS:
Overall Officials: Vesal Khalid, M.D., Study Chair — Northern Orthopaedic Department, Aalborg University Hospital, Denmark; Nils Johannesen, M.D., Study Chair — Cardiology Department, Aalborg University Hospital, Denmark
Locations (1):
- Northern Orthopaedic Division, Aalborg University Hospital,, Aalborg, Denmark